CLINICAL TRIAL: NCT06031415
Title: A Multicenter, Randomized, Placebo-Controlled Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of Multiple Ascending Doses of GS-0272 in Adult Participants With Rheumatoid Arthritis
Brief Title: Study of GS-0272 in Participants With Rheumatoid Arthritis
Acronym: MARASLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-666-6692
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Rheumatoid Arthritis (RA) Cohorts: GS-0272 or Placebo (Experimental): Part A will include participants with RA. Part A will have 3 cohorts. Each cohort in Part A will be randomized in a 3:1 ratio to receive either ascending doses of GS-0272 or placebo for 12 weeks.
  Dosing will begin in Cohort 1. Cohorts 2 and 3 will be initiated upon review of blinded safety data from the preceding cohort.
  Interventions: Drug: GS-0272; Drug: Placebo
- Part B: Active RA Cohort: GS-0272 or Placebo (Experimental): Part B will include participants with moderate-to-severe RA. Part B will have only 1 cohort (Cohort 4). Participants in Cohort 4 will be randomized in a 2:1 ratio to receive either GS-0272 or placebo for 12 weeks.
  Interventions: Drug: GS-0272; Drug: Placebo

INTERVENTIONS:
Drug: GS-0272 — Administered subcutaneously (for Part A) Administered intravenously or subcutaneously (for Part B)
Drug: Placebo — Administered subcutaneously (for Part A) Administered intravenously or subcutaneously (for Part B)

SUMMARY:
The goals of this clinical study are to learn more about the study drug, GS-0272, and its safety and tolerability following multiple doses in participants with rheumatoid arthritis (RA).

The primary objectives of this study are to assess the safety and tolerability of multiple ascending doses of GS-0272 and to characterize the pharmacokinetics of GS-0272 following multiple doses of GS-0272, in participants with RA.

ELIGIBILITY:
Key Inclusion Criteria:

* Age limit for the Republic of Korea for male or nonpregnant female is between 19 and 75 years of age.

Part A (Rheumatoid Arthritis (RA) Cohorts)-Specific Inclusion Criteria:

* Diagnosis of RA at least 3 months prior to screening fulfilling the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria.
* Ongoing treatment with 1 or 2 conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) for at least 12 weeks prior to the first dose of study drug, with a stable dose for at least 4 weeks prior to the first dose of study drug, as follows:
* Individuals must not be on a biologic disease-modifying antirheumatic drugs (bDMARD)/targeted synthetic disease-modifying antirheumatic drug (tsDMARD) at Day 1 or during the study and must discontinue b/tsDMARD use for at least 4 weeks (with the exception of rituximab, which must be discontinued for at least 16 weeks) prior to the first dose of study drug.

Part B (Active RA Cohort)-Specific Inclusion Criteria:

* Participant is seropositive as demonstrated by a positive anti-cyclic citrullinated peptide (anti-CCP) antibody and/or positive rheumatoid factor at screening.
* Participant has an elevated high-sensitivity C-reactive protein (hsCRP) greater than upper limit of normal (ULN).
* Participant has 6 or more swollen and 6 or more tender joints as assessed on the SJC66/TJC68. Distal interphalangeal joints will not be counted towards the 6 joint eligibility.
* Participant has had inadequate response or intolerance to at least 1 but not more than 3 bDMARD/tsDMARD therapeutics with no more than 2 MOAs. A lack of response is defined as documented continued or recurrent disease activity after at least 12 weeks of treatment of RA.

Key Exclusion Criteria:

* Meet any of the protocol-specified infection criteria (hepatitis C, Hepatitis B, HIV, tuberculosis, others).
* Inadequate response or intolerance to more than 3 bDMARDs/tsDMARDs with more than 2 MOAs.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Adverse Events (AEs) | First dose up to Week 12 plus 70 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) | First dose up to Week 12 plus 70 days
Percentage of Participants With Laboratory Abnormalities | First dose up to Week 12 plus 70 days
Pharmacokinetics (PK) of GS-0272: AUCtau | Day 1 predose through Day 197
  AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
PK of GS-0272: Cmax | Day 1 predose through Day 197
  Cmax is defined the maximum observed plasma drug concentration.
PK of GS-0272: Tmax | Day 1 predose through Day 197
  Tmax is defined as the time to maximum observed concentration.

SECONDARY OUTCOMES:
Prevalence of Antidrug Antibodies (ADAs) for GS-0272 | Baseline (Day 1) through Day 197
  Prevalence of ADAs will be measured as the proportion of participants who had at least one positive ADA sample (baseline or post-baseline) among all participants evaluable for ADA prevalence.
Incidence of ADAs for GS-0272 | Baseline (Day 1) through Day 197
  ADA incidence will be measured as the proportion of participants who have treatment-emergent ADA sample (post-baseline) among all participants evaluable for ADA incidence.
Part B: Change from Baseline in Disease Activity Score 28 (DAS28) C-Reactive Protein (CRP) in Participants with Moderate-to-Severe RA | Baseline, Week 12
  Disease Activity Score 28 C-Reactive Protein (DAS28 (CRP)) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), participant's global assessment of disease activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity) and CRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (24):
- United States (14):
  - Arizona Arthritis & Rheumatology Associates P.C., Glendale, California
  - Stanford School of Medicine, Division of Immunology & Rheumatology, Palo Alto, California
  - 1238 E. Arrow Hwy, Upland, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Greater Chicago Specialty Physicians/ Clinical Investigation Specialists, Niles, Illinois
  - Greater Chicago Specialty Physicians/Clinical Investigation Specialists, Inc., Schaumburg, Illinois
  - Summit Headlands LLC, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - PA Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Precision Comprehensive Clinical Research Solutions, Irving, Texas
  - 1600 Republic Parkway, Mesquite, Texas
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- IMSP Republican Clinical Hospital "Timofei Mosneaga", ARENSIA E.M., Chisinau, Moldova
- South Korea (3):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- United Kingdom (5):
  - Cambridge Clinical Research Centre, Rheumatology Research Unit - E6, Addenbrookes Hospital, Cambridge
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Kings College Hospital, London
  - Simbec Research Limited, Merthyr Tydfil
  - NIHR Wellcome Trust Clinical Research Facility, University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06031415